CLINICAL TRIAL: NCT04134013
Title: Nutrition Plus Chiropractic Care for Low Back Pain: a Randomized Clinical Trial
Brief Title: Nutrient Nutritional Advise for Low Back Pain Patients Seeking Chiropractic Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Parker University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Parker19_04
Record Dates: First submitted 2019-10-16; First posted 2019-10-21 (Actual); Last update posted 2022-01-14 (Actual); Status verified 2021-06

CONDITIONS: Low Back Pain; Nutrition Poor
Keywords: Chiropractic manipulation; spinal manipulation therapy; osteopathic manipulation
MeSH Terms: conditions — Low Back Pain; Malnutrition | interventions — Manipulation, Chiropractic

STUDY DESIGN:
Intervention Model Description: Participants will be randomized into one of two arms: 1) nutrition+chiropractic or 2) chiropractic only
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Project manager, participants, and investigator will be blinded to study. The registered dietitian will not be blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nutrition and Chiropractic (Experimental): LBP chiropractic adjustment per protocol and 4 Nutrient offerings (Vitamin Booster, Shake + 2 other offerings)
  Interventions: Dietary Supplement: Combination: Nutrition AND Chiropractic Adjustment
- Chiropractic Adjustment ONLY (Active Comparator): LBP chiropractic adjustment per protocol
  Interventions: Other: Chiropractic Adjustment: Spinal Manipulation Therapy

INTERVENTIONS:
Dietary Supplement: Combination: Nutrition AND Chiropractic Adjustment — LBP chiropractic adjustment per protocol, nutrition counseling/ 4 Nutrient offerings (Vitamin Booster, Shake + 2 other offerings)
  Arms: Nutrition and Chiropractic
Other: Chiropractic Adjustment: Spinal Manipulation Therapy — LBP chiropractic adjustment per protocol
  Arms: Chiropractic Adjustment ONLY

SUMMARY:
The nutritional intervention will reduce LBP and cause 10% weight loss.

DETAILED DESCRIPTION:
This feasibility study will assess a two-armed low-back pain (LBP) randomized, prospective clinical trial with nutritional offerings provided for one-arm.

ELIGIBILITY:
Inclusion Criteria:

BMI 25-40, Experiencing LBP (VAS>4, mechanical, chronic), not pregnant

Exclusion Criteria:

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2019-10-14 (Actual); Primary Completion 2019-11-23 (Actual); Study Completion 2020-11-26 (Actual)

PRIMARY OUTCOMES:
Low back pain evaluation using NPRS | Maximum six weeks of care
  Reduces Low Back Pain
Weight loss being measured using scale in pounds | Beginning of study and re-evaluation at the end of six weeks.
  Promotes weight loss

CONTACTS AND LOCATIONS:
Locations (1):
- Katie Pohlman, Plano, Texas, United States

REFERENCES:
- See also: Nutrient Foods — https://nutrientfoods.com/